CLINICAL TRIAL: NCT05128240
Title: A Randomised, Two-armed, Double-blinded Nutritional Study of Fish Oil on Skin Quality in Healthy Women
Brief Title: Nutritional Study of Fish Oil in Skin Quality in Healthy Women
Acronym: OPTIHUD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Epax Norway AS (Industry)
Collaborators: Møreforsking AS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P237921
Record Dates: First submitted 2021-11-04; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Skin Health
Keywords: skin; inflammation; wrinkles; trans epithelial water loss; fish oil; LCMUFA
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Placebo controlled, double blind intervention study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Interventions are given as 1g bovine capsules of equal size, weight and appearance, and provided in identical bottles with a coded label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 4x1g corn oil capsules
  Interventions: Dietary Supplement: Placebo
- Ceto 10 (Experimental): 4x1g capsules containing containing broad spectrum marine oil from north atlantic fish
  Interventions: Dietary Supplement: Ceto 10

INTERVENTIONS:
Dietary Supplement: Placebo — 1g corn oil capsules
  Arms: Placebo
Dietary Supplement: Ceto 10 — 1g capsules containing oil broad spectrum marine oil from north atlantic fish
  Arms: Ceto 10

SUMMARY:
The skin acts as a barrier against the external environment and prevents water loss from the body. Aging is a natural process leading to changes in the skin and fish oil has been shown to prevent inflammation, hyperpigmentation and UV-damage. This pilot study will determine skin characteristics after intervention with north atlantic fish oil.

DETAILED DESCRIPTION:
Women will be recruited to a placebo or fish oil group and be examined at pre- and post for skin quality parameters such as wrinkles, fine lines and trans-epithelial water loss.

ELIGIBILITY:
Inclusion Criteria:

Healthy women in the age of 30-65

Able to follow the following dietary restriction for 4 months (4 weeks wash-out, 3 months intervention):

* Do not take omega-3 supplements
* do not take supplements containing vitamin A
* do not take supplements containing collagen
* try to avoid using skin products containing vitamin A
* do not undergo skin treatment

Exclusion Criteria:

Pregnancy or breast feeding known allergy to seafood skin treatment the last 6 months planned skin treatment during the study period

-

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participation is based on self-assessment of gender identity
Enrollment: 30 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Determine the change in skin quality of healthy women after supplementation with fish oil compared to corn oil | 3 months
  Changes in quantitative analysis of facial inflammation, wrinkles and fine lines and skin texture will be performed using the VISIA Skin Analysis system. Measurements will be made at baseline and at end of supplementation period.

SECONDARY OUTCOMES:
Determine the change in omega-3 index (%EPA and DHA in red blood cells) after daily intake of 4g of north atlantic fish oil compared to placebo | 3 months
  Fatty acid profiles will be measured from blood samples using the Omega-quant test

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Midtbø, PhD, Principal Investigator — Møreforsking AS
Locations (1):
- Møreforsking AS, Ålesund, Norway

IPD SHARING:
Plan to Share IPD: No
Data will be presented as collective statistical data. Individual participant data may be shared on request, or if demanded by journals